CLINICAL TRIAL: NCT01298271
Title: Primary Prevention of Gastric Variceal Bleeding : Endoscopic Treatment Versus Non-selective Beta-blocker
Brief Title: A Randomized Trial of GVS Alone vs. Propranolol
Acronym: P-GVO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSC99-2314-B-010-049-MY3
Record Dates: First submitted 2010-10-04; First posted 2011-02-17 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Bleeding Gastric Varices; Liver Cirrhosis
Keywords: gastric variceal bleeding; primaryprevention; cyanoacrylate injection; non-selective beta-blocker
MeSH Terms: conditions — Liver Cirrhosis | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyanoacrylate (No Intervention): Endoscopic Cyanoacrylate Injection treatment of primary prevention GVB
- Propranolol (Active Comparator): Propranolol is used for primary prevention of GVB
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — Starting from 20 mg daily, titrated weekly to decrease heart rate more than 25 % of baseline, administrated during the whole study period
  Other Names: Inderal, Cardolol
  Arms: Propranolol

SUMMARY:
Design a randomized trial to compare the effect of endoscopic cyanoacrylate injection obliteration versus non-selective beta-blocker in the primary prevention of gastric variceal bleeding.

DETAILED DESCRIPTION:
Up to date, the treatment of gastric variceal bleeding (GVB) is still sub-optimal in contrast to the treatment of esophageal variceal bleeding (EVB), which already had a big improvement of prognosis in recent two decades. Gastric varices (GV) rarely rupture. However should it occur, the outcome would be worse than rupture of esophageal varies (EV). Rupture of GV is characteristic of a higher rebleeding rate (90%), a requirement for a larger amount of blood transfusion and a higher mortality (40-50%). Therefore, primary prevention of GV rupture is critically important. The management of GV has been focused on treatment of acute GVB. Tissue adhesive (cyanoacrylate) may polymerize and occlude the vascular channels in seconds and obliterate for more than 70% cases of GV. The rebleeding rate after endoscopic cyanoacrylate injection(GVO) of acute GVB is around 30~40% and expertise is required to reduce the embolic complications and instrumental injuries.GVO may arrest more than 90% active GVB. The 2005 Baveno IV International Consensus and 2007 AASLD Guidelines endorsed that endoscopic cyanoacrylate injection is the first line treatment for acute GVB. However, its efficacy on prevention of first GV bleeding is not known. Non-selective beta-blocker (NSBB) is effective to prevent first and second bleeding from esophageal varices. The 2005 Baveno IV International Consensus and 2007 AASLD Guidelines also endorsed that NSBB is the first choice for the primary prevention of EVB. However, its effect on gastric variceal hemorrhage has never been clarified. Actually, GV usually has a large gastrorenal shunting and the portal pressure of GV is lower than that of EV. For ethical concerns, NSBB is usually be used for primary prevention of GVB, the preventive effect of NSBB had never been proved. Study on the primary prevention of GVB is scanty. This is an important issue prompted by current portal hypertension experts. The investigators have a lot of experience in the treatment of gastric variceal bleeding and published fruitful results in high ranking journals. Therefore, the investigators design a randomized trial to compare the effect of endoscopic cyanoacrylate injection obliteration versus non-selective beta-blocker in the primary prevention of gastric variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. patients with live cirrhosis and/or hepatoma
2. Aged 18 to 80, who had endoscopy-Proven EV(-)GV(+)or EV<GV

Exclusion Criteria:

1. Patients had previous endoscopic, surgical treatment or Transjugular Intrahepatic Portosystemic Shunt
2. Had a terminal illness of any major organ system,such as heart failure, kindey failure,COPD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | 3 year

SECONDARY OUTCOMES:
complication surivial | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Hou, MD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Veteran General Hospital-Taipei, Taipei, Taiwan